CLINICAL TRIAL: NCT07023081
Title: A PHASE 1, OPEN-LABEL STUDY TO EVALUATE THE SAFETY AND TOLERABILITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY CHINESE ADULTS, CHILDREN, AND INFANTS
Brief Title: A Study to Understand the Safety of the 20vPnC Vaccine in Healthy Chinese Adults, Children, and Infant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B7471021
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Masking Description: This is an open label study. Participant, investigators, and sponsor will be unblinded to the participant's assigned study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1 (Experimental): Participants will receive 1 dose of 20vPnC Vaccine.
  Interventions: Biological: 20vPnC
- Cohort 2 (Experimental): Participants will receive 1 dose of 20vPnC Vaccine.
  Interventions: Biological: 20vPnC
- Cohort 3 (Experimental): Participants will receive 2 doses of 20vPnC Vaccine on Day 1 (Vaccination 1) and 56 to 70 days after Vaccination 1 (Vaccination 2).
  Interventions: Biological: 20vPnC
- Cohort 4 (Experimental): Participants will receive 3 doses of 20vPnC Vaccine on Day 1 (Vaccination 1), 28 to 56 days after Vaccination 1 (Vaccination 2), and at 365 to <455 days of age and at least 56 days after Vaccination 2 (Vaccination 3).
  Interventions: Biological: 20vPnC
- Cohort 5 (Experimental): Participants will receive 4 doses of 20vPnC Vaccine on Day 1 (Vaccination 1), 42 to 63 days after Vaccination 1 (Vaccination 2), 42 to 63 days after Vaccination 2 (Vaccination 3), and at 365 to <455 days of age (Vaccination 4).
  Interventions: Biological: 20vPnC
- Cohort 6 (20vPnC) (Experimental): Participants will receive 4 doses of 20vPnC Vaccine on Day 1 (Vaccination 1), 42 to 63 days after Vaccination 1 (Vaccination 2), 42 to 63 days after Vaccination 2 (Vaccination 3), and at 365 to <455 days of age (Vaccination 4).
  Interventions: Biological: 20vPnC
- Cohort 6 (13vPnC) (Active Comparator): Participants will receive 4 doses of 13vPnC Vaccine on Day 1 (Vaccination 1), 42 to 63 days after Vaccination 1 (Vaccination 2), 42 to 63 days after Vaccination 2 (Vaccination 3), and at 365 to <455 days of age (Vaccination 4).
  Interventions: Biological: 13vPnC

INTERVENTIONS:
Biological: 20vPnC — 20vPnC vaccine
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6 (20vPnC)
Biological: 13vPnC — 13vPnC vaccine
  Arms: Cohort 6 (13vPnC)

SUMMARY:
The purpose of this study is to learn about the safety of the 20-valent pneumococcal conjugate vaccine (20vPnC) among adults, children, and infants, as well as the immunogenicity of 20vPnC among infants and children under 2 years of age in China. This vaccine will be given as per the age-specific dosing schedules among healthy adults, children and infants in China.

This study is seeking healthy participants of 6 groups:

* Group 1: Adults ≥18 to <50 years of age
* Group 2: Children ≥2 to <6 years of age
* Group 3: Children ≥12 months to <2 years of age
* Group 4: Infants ≥7 to <12 months of age
* Group 5: Infants ≥42 to ≤98 days of age
* Group 6: Infants ≥42 to ≤98 days of age

All participants in Group 1 to 5, in this study will receive 20vPnC as per the age-specific dosing schedules:

* Group 1: participants will receive 1 dose of 20vPnC.
* Group 2: participants will receive 1 dose of 20vPnC.
* Group 3: participants will receive 2 doses of 20vPnC. Dose 2 will be given 56 to 70 days after Dose 1.
* Group 4: participants will receive 3 doses of 20vPnC. Dose 2 will be given 28 to 56 days after Dose 1, and Dose 3 will be given at 365 to <455 days of age and at least 56 days after Dose 2.
* Group 5: participants will receive 4 doses of 20vPnC. Dose 2 will be given 42 to 63 days after Dose 1, and Dose 3 should be given 42 to 63 days after Dose 2, and Dose 4 should be given at 365 to <455 days of age.

Participants in Group 6 will be randomized in a 1:1 ratio to received either 20vPnC or 13vPnC:

- Group 6: participants will receive 4 doses of 20vPnC or 13vPnC. Dose 2 will be given 42 to 63 days after Dose 1, and Dose 3 should be given 42 to 63 days after Dose 2, and Dose 4 should be given at 365 to <455 days of age.

The study will look at the experiences of people receiving the study vaccine. The study will also look at the immune response of some people receiving the study vaccine. This will help decide if the study vaccine is safe.

The total duration of taking part in the study from each group is:

* Participants in Group 1 and Group 2 will take part for about 6 months, with 6 visits.
* Participants in Group 3 will take part for about 8 months, with 9 visits.
* Participants in Group 4 will take part for about 12 months, with 8 visits.
* Participants in Group 5 and 6 will take part for about 16 to 19 months, with 11 visits.

ELIGIBILITY:
Key inclusion criteria:

* Male or female participants:

  * Adults ≥18 to <50 years of age
  * Children ≥2 to <6 years of age
  * Children ≥12 months to <2 years of age
  * Infants ≥7 to <12 months of age
  * Infants ≥42 to ≤98 days of age
* Healthy participants determined by clinical assessment and clinical judgment, to be eligible for the study.

Key exclusion criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention, or any diphtheria toxoid-containing vaccine.
* History of microbiologically proven invasive disease caused by S pneumoniae.
* Congenital, functional, or surgical asplenia.
* Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt during study participation.
* Determined as not eligible by the investigator based on the participant's past and present health condition(s), medication(s) and treatment(s).

Please refer to the study contact for further eligibility details.

Ages: 42 Days to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2027-05-14 (Estimated); Study Completion 2027-05-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting prespecified local reactions within 7 days following each study intervention | Within 7 days of each study intervention
  Prespecified local reactions following each study intervention
Percentage of participants reporting prespecified systemic events within 7 days following each study intervention | Within 7 days of each study intervention
  Prespecified systemic events following each study intervention
Percentage of participants reporting adverse events (AEs) from the first study intervention through 1 month following the last study intervention administration | 1 month after the last vaccination
  AEs occurring through 1 month following the last study intervention administration for participants of adults ≥18 to <50 years of age at the time of consent, and children and infants ≥7 months to <6 years of age at the time of consent.
Percentage of participants reporting AEs from the first study intervention through 1 month following the third study intervention. | From the first study intervention to 1 month after the third study intervention
  AEs occurring from the first study intervention through 1 month following the third study intervention in infants ≥42 to ≤98 days of age at the time of consent.
Percentage of participants reporting AEs from the fourth study intervention to 1 month following the fourth study intervention. | From the fourth study intervention to 1 month after the fourth study intervention
  AEs occurring from the fourth study intervention to 1 month following the fourth study intervention in infants ≥42 to ≤98 days of age at the time of consent.
Percentage of participants reporting serious adverse events (SAEs) throughout the study | From the first study intervention to 6 months after the last study intervention
  SAEs through 6 months following last study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Nanning, Guangxi
  - Wuming District Center for Disease Control and Prevention, Chengxiang, Nanning

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471021